CLINICAL TRIAL: NCT00019331
Title: Vaccine Therapy With Tumor Specific Mutated Ras Peptides and IL-2 or GM-CSF for Adult Patients With Solid Tumors
Brief Title: Vaccine Therapy Plus Biological Therapy in Treating Adults With Metastatic Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065656; NCI-97-C-0141F; NCI-T96-0078; NCT00001581 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2004-04

CONDITIONS: Colorectal Cancer; Endometrial Cancer; Head and Neck Cancer; Liver Cancer; Lung Cancer; Melanoma (Skin); Pancreatic Cancer; Testicular Germ Cell Tumor; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV colon cancer; recurrent non-small cell lung cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; recurrent colon cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; stage IV endometrial carcinoma; recurrent endometrial carcinoma; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; stage IV papillary thyroid cancer; stage IV follicular thyroid cancer; thyroid gland medullary carcinoma; anaplastic thyroid cancer; recurrent thyroid cancer; stage IV melanoma; recurrent melanoma; stage IV non-small cell lung cancer; unspecified adult solid tumor, protocol specific; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; adult primary hepatocellular carcinoma; pulmonary carcinoid tumor; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; insular thyroid cancer; recurrent salivary gland cancer; stage IV salivary gland cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Colorectal Neoplasms; Endometrial Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Lung Neoplasms; Melanoma; Pancreatic Neoplasms; Testicular Germ Cell Tumor; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Hepatocellular; Testicular Neoplasms; Thyroid Cancer, Papillary; Adenocarcinoma, Follicular; Carcinoma, Medullary; Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — aldesleukin; sargramostim

INTERVENTIONS:
Biological: aldesleukin
Biological: ras peptide cancer vaccine
Biological: sargramostim
Drug: DetoxPC

SUMMARY:
RATIONALE: Vaccines made from a peptide may make the body build an immune response to kill tumor cells. Combining vaccine therapy with interleukin-2 and/or sargramostim may be a more effective treatment for solid tumors.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy plus interleukin-2 and/or sargramostim in treating adults who have metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether endogenous cellular immunity to a tumor-specific mutated ras protein is present in cancer patients.
* Determine whether vaccination with synthetic peptides corresponding to the tumor's ras mutation with DetoxPC adjuvant, interleukin-2 (IL-2), and/or sargramostim (GM-CSF) can induce or boost a patient's cellular immunity to that particular mutation.
* Determine the type and characteristics of the cellular immune response generated.
* Determine the tolerance to and toxicity spectrum of such peptides given with DetoxPC adjuvant along with IL-2 and/or GM-CSF.
* Correlate immune response with tumor response in patients treated with these regimens.

OUTLINE: Patients are assigned to one of three treatment groups.

* Group I (closed to accrual 6/4/01): Patients receive tumor-specific ras peptide vaccine with DetoxPC subcutaneously (SC) once every 5 weeks for 3 courses. Beginning 4 days after vaccination, patients receive interleukin-2 (IL-2) SC 5 days a week for 2 weeks.
* Group II (closed to accrual 6/4/01): Patients receive sargramostim (GM-CSF) SC daily beginning 1 day prior to the vaccination and continuing for 4 days. Patients receive the vaccination as in group I immediately followed by GM-CSF on day 2. Patients are vaccinated once every 4 weeks for 3 courses.
* Group III: Patients receive the vaccination and IL-2 as in group I and GM-CSF as in group II.

In all groups, patients receive up to 15 vaccinations in the absence of disease progression.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A maximum of 60 patients (20 per treatment group) will be accrued for this study within 2-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumors potentially expressing mutant ras, including colon, lung, pancreas, thyroid, endometrial, head and neck, testicular, hepatocellular, and melanoma
* Ras mutations must be one of the following point mutations at codon 12:

  * Glycine to cysteine
  * Glycine to aspartic acid
  * Glycine to valine
* Metastatic disease for which no known chemotherapy or radiotherapy would increase survival
* Tumor tissue must be available for determination of ras mutation
* No prior CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT/SGPT no greater than 4 times normal
* No hepatitis B or C infection

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No active ischemic heart disease (New York Heart Association class III or IV)
* No myocardial infarction within the past 6 months
* No history of congestive heart failure, ventricular arrhythmias, or other arrhythmias requiring therapy

Immunologic:

* No prior allergy to eggs
* No prior autoimmune disease, including the following:

  * Autoimmune neutropenia, thrombocytopenia, or hemolytic anemia
  * Systemic lupus erythematosus, Sjogren's syndrome, or scleroderma
  * Myasthenia gravis
  * Goodpasture syndrome
  * Addison's disease, Hashimoto's thyroiditis, or active Graves' disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other active malignancy except curatively treated carcinoma in situ of the cervix or basal cell skin cancer
* No active infection requiring antibiotics
* No medical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* At least 4 weeks since prior steroids and recovered

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-10; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry L. Gause, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States